CLINICAL TRIAL: NCT06618586
Title: Get Social Media and Risk-Reduction Training (GET SMART)
Brief Title: Get Social Media and Risk-Reduction Training
Acronym: GETSMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Washington University School of Medicine (Other); Boston Medical Center (Other); Boston University (Other); University of Massachusetts, Worcester (Other); Columbia University (Other); University of Colorado, Denver (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Rachel Moon, MD, Professor, Department of Pediatrics, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 202401227; R01HD110568-01A1 (NIH)
Record Dates: First submitted 2024-08-27; First posted 2024-10-01 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Infant Death; Sudden Infant Death
Keywords: Safe Sleep; Mobile Messaging
MeSH Terms: conditions — Infant Death; Sudden Infant Death

STUDY DESIGN:
Intervention Model Description: This is a hybrid type 3 implementation-effectiveness cluster randomized trial at 20 US birth hospitals. In a crossover design separated by a 1-month washout period, we will test 2 strategies for recruitment of mothers into the 2-month-long TodaysBaby mobile safe sleep education program: 1) The original TodaysBaby implementation strategy (HT), in which hospital staff recruit mothers and view the first 2 videos with them; and 2) A new low-touch (LT) hospital implementation strategy, in which mothers are attracted to TodaysBaby through direct-to-consumer marketing and sign themselves up using a QR code.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- New low touch (LT) hospital implementation strategy (Experimental): This will occur during either the first or second 6-month intervention time period (order randomly assigned). For the period of time hospitals are randomized into this arm mothers will be attracted to TodaysBaby through direct-to-consumer marketing and sign themselves up using a QR code. These mothers will also receive standard postpartum care.
  Interventions: Behavioral: TodaysBaby
- Original high touch (HT) hospital implementation strategy (Active Comparator): This will occur during either the first or second 6-month intervention time period (order randomly assigned). For the period of time hospitals are randomized into this arm hospital staff will help mothers sign up and view the first 2 TodaysBaby in a one-on-one conversation format. These mothers will also receive standard postpartum care.
  Interventions: Behavioral: TodaysBaby
- Control- Standard of Care (No Intervention): During the 3 months immediately prior to the first intervention time period, hospitals will recruit approximately 100 mothers to complete surveys regarding infant care practices. These mothers will also receive postpartum standard of care.

INTERVENTIONS:
Behavioral: TodaysBaby — The TodaysBaby intervention is comprised of: 1) Text message-delivered, short educational videos in the first 2 months after birth, with each video timed to match content addressing anticipated barriers and facilitators to adhering to guidelines (e.g. parental concerns that infant will choke while supine). Participants will also have access to a web portal where intervention videos will be maintained. 2) Text queries regarding safe sleep practices, which collect data on sleep practices in near real-time and provide reinforcement of adherence. Mothers will receive 1-2 text message questions weekly that assess sleep practices in near real-time .
  Arms: New low touch (LT) hospital implementation strategy; Original high touch (HT) hospital implementation strategy

SUMMARY:
This study examines the implementation of the TodaysBaby™ mobile safe sleep intervention program in US hospitals. The main aims of this study are to examine: 1) differences in program penetration and the equity of penetration according to income and race/ethnicity; 2) differences in feasibility, acceptability, sustainability and fidelity top the intervention; and 3) the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must speak English or Spanish
* Must live in the United States
* Must have given birth to a healthy, term infants (37 weeks or greater) and be discharged within 7 days of birth
* Must plan to care for infant and live in the same household as infant after birth
* Must enroll in the TodaysBaby program by the time their infant is 7 days of age

Exclusion Criteria:

* A prenatal diagnosis expected to have impact on infant care practices not compatible with study goals, such as supine infant sleep positioning.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Penetration of sign up for TodaysBaby | First week after birth
  Rate of sign up for TodaysBaby among mothers that sign up during the different implementation strategies
Equity of sign up for TodaysBaby | First week after birth
  Differences in rate of sign up for TodaysBaby by maternal insurance status and race/ethnicity among mothers that sign up during different implementation strategies

SECONDARY OUTCOMES:
Feasibility of implementation | Within a year of participant enrollment (qualitative) and >60 day after birth survey
  Staff perception that the implementation strategies were successfully used or carried out (measured through semi-structured interviews; Rate of maternal report that signing up for TodaysBaby was simple and fast
Acceptability | Within a year of participant enrollment
  Staff perception that the delivery of the implementation strategies was satisfactory (measured through semi-structured interviews)
Sustainability | Within a year of participant enrollment (qualitative) and during the 6-month study implementation periods
  Staff perception that the implementation strategies could continue to be delivered after the end of the study (measured through semi-structured interviews); monthly penetration rates
Fidelity | First 60 days after birth
  Number of videos viewed by mother, divided by total videos among mothers enrolled in the different implementation strategies
Effectiveness of TodaysBaby on safe sleep practices | 60-180 days (average 80 days) after birth survey
  We will measure 4 sleep practices in the past 2 weeks among mothers enrolled in the different implementation strategies:
  Sleep position: % reporting supine position only Sleep location: % reporting roomsharing not bedsharing only Soft bedding: % reporting no soft bedding in sleep space Pacifier: % reporting usual pacifier use when infant sleeping
Program cost of TodaysBaby | 60-180 days during the program sign up periods.
  Differences in rate of sign up for TodaysBaby by maternal insurance status and race/ethnicity among mothers that sign up during different implementation strategies

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Y Moon, MD, Principal Investigator — University of Virginia School of Medicine
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No